CLINICAL TRIAL: NCT00162721
Title: Phase III Study About the Effects of the Addition of Polychemotherapy to Adjuvant Radiotherapy in the Treatment of Non-Metastatic Uterine Sarcomas
Brief Title: The Addition of Polychemotherapy to Adjuvant Radiotherapy in the Treatment of Non-Metastatic Uterine Sarcomas
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SARC-GYN1
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-08

CONDITIONS: Uterine Sarcoma
Keywords: Uterine sarcoma non metastatic
MeSH Terms: interventions — Doxorubicin; Ifosfamide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: doxorubicin, ifosfamide, cisplatin

SUMMARY:
This is a Phase III study about the effects of the addition of polychemotherapy to adjuvant radiotherapy in the treatment of non-metastatic uterine sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed uterine sarcoma (rereading in reference centers)
* Leiomyosarcoma, adenosarcoma, carcinosarcoma and high grade endometrial stromal sarcoma
* All stages <= stage III (FIGO modified for endometrial carcinoma)
* Full surgical exeresis
* Age >= 18 years and physiological age <= 65 years
* Negative extension check-up (thoracic and abdomino-pelvic TDM)
* Performance status (PS) <= 2 (ECOG)
* Normal haematologic functions (absolute neutrophil count > 1,500/mm3, platelets > 100,000/mm3)
* Serum creatinine < 1.25 x ULN
* Good hepatic check-up (total serum bilirubin < 1.5 x ULN; AST or ALT < 2.5 x ULN)
* Absence of neuropathy > grade 1
* Left ventricular ejection fraction > 50% (by isotopic or ultrasound scan determination)
* Written informed consent

Exclusion Criteria:

* Low grade endometrial stromal sarcoma
* Time since surgery > 8 weeks
* Specific contraindications to the studied treatment (cardiac, kidney, or hepatic ones)
* Antecedents or evolutive psychiatric disorder
* Concurrent active infection or other serious uncontrolled systemic disease
* Antecedents of cancer but a cutaneous basocellular one or an in situ epithelioma of the cervix

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2001-09

PRIMARY OUTCOMES:
Effects of the addition of an adjuvant chemotherapy to adjuvant pelvic radiotherapy on a 3 year event-free survival in the treatment of localized uterine sarcomas

SECONDARY OUTCOMES:
Effects of the addition of an adjuvant chemotherapy to adjuvant pelvic radiotherapy on overall survival
Evaluation of global toxicity of the treatment in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Pautier, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France